CLINICAL TRIAL: NCT03014986
Title: Current Treatment of HCV Infection After HSCT
Status: Completed | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: (4)8414107
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C
Keywords: HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients who receive HCV treatment: HSCT patients with HCV who are receiving (or has recently received) HCV treatment
- Patients who do not receive HCV treatment: HSCT patients with HCV who have not received treatment

SUMMARY:
The availability of novel therapies with DAAs might prompt clinicians caring for HSCT recipients with HCV infection to prescribe the treatment more frequently and possibly earlier after HSCT. Since numerous possible therapeutic combinations exist, the choice of the most appropriate one is not straightforward. It depends not only on its efficacy, toxicity and rate of pharmacological interactions, but also on availability (both through healthcare system and in expanded access programs), and cost.

This observational prospective study will focus on treatment strategies in HSCT recipients with HCV infection. The main focus will be the therapeutic approach, the combination of drugs chosen, the length of treatment and the outcome. The main reasons for treating or not treating HSCT recipients with HCV infection will be also explored. Compared to previous cohorts, this study might provide additional data in the area of non-invasive assessment of fibrosis, HCV-RNA levels and genotyping.

In order to get as much data as possible on HCV treatment, patients with chronic HCV infection transplanted during the last 10 years will be included.

Finally the prevalence of HCV-RNA positive patients among those transplanted in the year 2016 will be reported.

DETAILED DESCRIPTION:
Introduction:

According to previous EBMT studies, approximately 6% of HSCT recipients were HCV-positive (Locasciulli et al. Transplantation 1999). Despite the fact that HSCT recipients with chronic HCV infection are prone to HCV-morbidity (end stage liver disease, hepatocellular carcinoma, the need for liver transplant), only about half (44% and 61%) of long term survivors of HSCT were offered specific treatment (Ljungman et al. BMT 2012; Peffault de Latour et al. BMT 2005). The median time from HSCT to treatment was long and the efficacy was far from satisfactory (approximately 50%) (Ljungman et al. BMT 2012). Since 2011 novel oral directly acting antiviral agents (DAA) have been developed and marketed. DAAs offer the advantage of higher efficacy, shorter duration and reduced treatment toxicity; together with the possibility of exclusively oral, interferon- or interferon/ribavirin-free regimens.

Short description of the study:

The availability of novel therapies with DAAs might prompt clinicians caring for HSCT recipients with HCV infection to prescribe the treatment more frequently and possibly earlier after HSCT. Since numerous possible therapeutic combinations exist, the choice of the most appropriate one is not straightforward. It depends not only on its efficacy, toxicity and rate of pharmacological interactions, but also on availability (both through healthcare system and in expanded access programs), and cost.

This observational prospective study will focus on treatment strategies in HSCT recipients with HCV infection. The main focus will be the therapeutic approach, the combination of drugs chosen, the length of treatment and the outcome. The main reasons for treating or not treating HSCT recipients with HCV infection will be also explored. Compared to previous cohorts, this study might provide additional data in the area of non-invasive assessment of fibrosis, HCV-RNA levels and genotyping.

In order to get as much data as possible on HCV treatment, patients with chronic HCV infection transplanted during the last 10 years will be included.

Finally the prevalence of HCV-RNA positive patients among those transplanted in the year 2016 will be reported.

Research design:

Over the period of 24 months, all HCV-RNA positive patients who received autologous or allogeneic transplant from any time to May 2017 and are followed at transplant centres will be enrolled.

Data regarding the patients who are receiving (or has recently received) HCV treatment (group 1) will be collected in Form 1 (FORM 1 - HCV TREATMENT) and 6 months after the end of treatment in Form 4 (FORM 4 - POST HCV TREATMENT FOLLOW UP FORM)

Data regarding the baseline characteristics of HCV-RNA positive patients who are not being treated (group 2) will be collected in Form 2 (FORM 2 - HCV-RNA positive patients - BASELINE) and then at the end of the recruitment period (December 2017 +/- 3 months) in Form 3 (FORM 3 - HCV-RNA positive patients - FOLLOW UP FORM).

If patients from group 2 start treatment, their data thereafter should be reported in Form 1 and then Form 4.

Including: Duration of the study Recruitment period (visits date for HCV-RNA+ patients) starts December 2015 till November 2017. All the patients will be followed for a minimum additional period of 6 months from the end of recruitment period.

Patients, in whom HCV treatment started before December 2015, will be also included if followed during the study period with the aim of establishing the efficacy of the recent HCV-treatment (HCV-RNA testing to establish SVR at 12 and 24 weeks after EOT).

Study Population:

All HCV-RNA positive patients transplanted from anytime until May 2017, followed from December 2015 to November 2017.

Data Collection & Statistical Analysis Plan:

All data collection will be performed by the IDWP Data Office (Leiden) according to EBMT guidelines.

Data from Med A + Med B with the following:

At the first visit occurring between January 2016 and December 2017:

* Date of diagnosis of HCV
* Quantitative HCV-RNA
* Genotype of HCV, IL28B polymorphism in case of G1 and G4
* Fibrosis according to elastography and/or biopsy (grade and date) and/or serological assays
* Previous anti-HCV treatment (date, type, duration, side-effects, outcome)
* HBV status (chronic active infection, chronic inactive infection, resolved infection, immunised) and HIV status
* Clinical data: ALT, albumin, PT, serum creatinine, encephalopathy, ascites, white cell count, Hb, platelets, dialysis, hepatocellular carcinoma (HCC)
* Concomitant pharmacological treatment
* Occurrence of VOD (grade, date)
* Acute or chronic GVHD (grade, date)

At the end of the study for not treated HCV-RNA- positive patients (December 2017, +/- 3 months):

* Quantitative HCV RNA (date)
* Fibrosis according to elastography and/or biopsy (grade and date) and/or serological assays
* Chronic GvHD (grade, date)
* Clinical data: ALT, albumin, PT, serum creatinine, encephalopathy, ascites, white cell count, Hb, platelets, dialysis
* Presence of hepatocellular carcinoma (HCC)
* Reason for treatment or reason for not starting HCV-treatment
* Reason for death, if applicable

In case of treatment:

* Treatment regimen (drugs, length)
* On treatment response (all HCV-RNA levels and dates)
* Concomitant pharmacological treatment
* SVR at 12 and 24 weeks after the end of treatment
* Reason for discontinuation (EOT, side tolerability, etc.)
* Treatment associated side effects (type, grade, its treatment, date of onset and date of resolution), including pharmacological interactions
* Treatment payment (national healthcare system, expanded access, research protocol, etc.)

Statistical analysis

Main outcome variables:

1. Description of treatment approach of HCV infection The type of treatment (drugs, doses) for HCV will be described. The following variables will be described in patients with and without treatment for HCV: age, type of transplant, type of underlying disease, status of the underlying disease, presence of relapse, time from HSCT (from Med A form); HCV-RNA level, grade of fibrosis, genotype, previous acute or chronic GVHD (grade max.), Child-Pugh score (to be calculated from clinical variables), presence of HCC.
2. SVR at week 12 and 24 after the EOT, yes/no The following variables will be described in patients with and without sustained viral response (SVR) at week 12 and 24 after the EOT: age, type of transplant, type of underlying disease, status of the underlying disease, presence of relapse, time from HSCT (from Med A form); HCV-RNA level, grade of fibrosis, genotype and polymorphism if applicable, previous acute or chronic GVHD (grade max.), Child- Pugh score (to be calculated from clinical variables), presence of HCC, type of treatment (particular regimen, interferon-free vs. interferon-based regimen, etc), toxicity, on treatment response, presence of possible interacting drugs.

Categorical variables to be compared according to chi-square test of exact Fisher's test if applicable, continuous variables to be compared with Mann-Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* HSCT recipients (allogeneic and autologous) with HCV infection
* Transplanted from anytime until May 2017, followed from December 2015 to November 2017.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All HCV-RNA positive patients transplanted from anytime until May 2017, followed from December 2015 to November 2017
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-12; Primary Completion 2020-03 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Description of treatment approach of HCV infection | 6 months
  The type of treatment (drugs, doses) for HCV will be described.

SECONDARY OUTCOMES:
SVR at week 12 and 24 after the EOT, yes/no | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simone Cesaro, Study Chair — Paediatric Haematology Oncology, Policlinico G.B. Rossi; Malgorzata Mikulska, Principal Investigator — University of Genoa, San Martino University Hospital
Locations (7):
- Centre Hospitalier de Meaux, Meaux, France
- Italy (4):
  - Ospedale San Raffaele s.r.l., Milan
  - Ospedale Santa Maria della Misericordia, Perugia
  - Ospedale Civile, Pescara
  - Policlinico G.B. Rossi, Verona
- Spain (2):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital de la Princesa, Madrid

IPD SHARING:
Plan to Share IPD: Undecided